CLINICAL TRIAL: NCT04478799
Title: Long Term Outcome of Transcutaneous Posterior Tibial Nerve Stimulation in Treatment of Functional Non-Retentive Fecal Incontinence
Brief Title: Transcutaneous Posterior Nerve Stimulation inTreatment of Fecal Incontience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Associate Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Banha University
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Fecal Incontinence
Keywords: Posterior Tibial Nerve Stimulation; Fecal Incontinence; Long Term Effect
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: The current single-blind randomized controlled study included 102 children with FNRF who were randomly allocated into two groups. Group 1, Bilateral transcutaneous posterior tibial nerve stimulation and group B, Sham TPTNS. Inclusion criteria included those with FI and normal defecation frequency, normal bowel habits and stool consistency. Children younger than 4 years or those who are not cooperative, or those with traumatic sphincter injury, fecal impaction, spinal diseases causing incontinence, anorectal malformation, were excluded from the study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Transcutanous Posterior Tibial Nerve Stimulation) (Experimental): Patients belonging to the group A received Transcautanoues posterior tibial nerve stimulation plus diet and Kegel exercises
  Interventions: Device: Transcutanous Posterior Tibial Nerve Stimulation
- Group B (Sham Control) (Sham Comparator): Patients belonging to the group B received Sham Transcautanoues posterior tibial nerve stimulation plus diet and Kegel exercises
  Interventions: Device: Sham Transcutanous Posterior Tibial Nerve Stimulation

INTERVENTIONS:
Device: Transcutanous Posterior Tibial Nerve Stimulation — children were managed by bilateral TPTNS following the procedure described in 2006 by Queralto et al(11). A positive auto-adhesive electrode was applied 1.5 inch above the medial malleolus over the S3 dermatome. A second negative electrode was applied just below the same malleolus. Electrical stimulation device (EMS physio Ltd, OX129 F, England) was connected to both electrodes. This device delivers a low frequency current (10 Hz), and the intensity was gradually increased till flexion of the big toe or spread out of the other toes in a fan shape occurred. Then the intensity was lowered to (10 Hz) again to avoid the motor response of the toes. Intensity was determined by the child's sensitivity. The procedure was done for 20-30 minutes and repeated2 times per week for 3 months
  Arms: Group A (Transcutanous Posterior Tibial Nerve Stimulation)
Device: Sham Transcutanous Posterior Tibial Nerve Stimulation — Sham transcutaneous stimulation Patients also had twice-weekly 20-30-min sessions for 3 months. The same self-adhesive electrodes as used for group A were employed, placed in a similar position. The stimulator was briefly switched on for 30 s to induce only a minor electrical sensation in the skin, and was then turned off for the rest of the treatment. This short duration was given for only for a few seconds to avoid lower limb stimulation. Patients in all TWO groups were told that they may or may not have any perception of the electrical stimulation. Without prior knowledge of what to expect from treatment, this enabled the sham group to act as a control. In order to improve on the blinding effect of the study, the electronic display window of the stimulators was shielded from the patients in the TWO groups. All patients underwent therapy in individual screened cubicles to prevent comparison between patients of the treatment being administered.
  Arms: Group B (Sham Control)

SUMMARY:
Shafik and colleagues were the first to report the use of posterior tibial nerve stimulation (PTNS) for FI, and they documented improved continence after 4 weeks course. Subsequent studies documented percutaneous and transcutaneous PTNS as effective methods for treatment of FI, with a short term reduction in incontinence episode by 50-80 %. Percutaneous PTNS (PPTNS) showed a greater effect than transcutaneous PTNS (TPTNS) and this may be assumed due to the presence of the stimulating electrode very close to the posterior tibial nerve. However, TPTNS is more preferable to percutaneous PTNS because of the concern about the insertion of a needle may result in stimulation that is sufficient to produce a neuromodulatory effect.

DETAILED DESCRIPTION:
Treatment of FNRFI is often difficult and requires prolonged therapies with unexpected responses and frequent relapses. The corner-stones in treatment of FNRFI are education, positive motivation, and toilet training. Preparation of children and their parents for a long-lasting treatment is mandatory with the expectation of many ups and downs. The main goal is to have regular bowel movements and normal continence and this can be achieved by teaching the child the importance of regular toilet use and avoid urges.

Many previous studies, reported the short term effect of TPTNS in treatment of FNRFI. However, there are sufficient studies evaluating the long term effect of TPNS and this has motivated the authors to conduct of this study The aim of this study is to evaluate the Long term outcome and quality of life in children with Functional non-retentive fecal incontinence and received Bilateral Transcutaneous posterior tibial nerve stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from (6-14 years) with FNRFI with normal bowel habits
* Children with normal defecation frequency and normal stool consistency
* Children with incontinence score ranging from 8-22 according to Vaizey score

Exclusion Criteria:

* Children who have traumatic sphincter injury.
* Children who have Fecal impaction
* Children who have Spinal diseases causing incontinence
* Children who have Anorectal malformation
* Children who were not cooperative

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Number of incontinence episodes | 24 months
  Change in the number of incontinence episodes
Incontinence Score using Vaizey incontinence score | 24 months
  Questionnaire ranging from zero (indicating complete continence) to 24 (indicating total incontinence).

SECONDARY OUTCOMES:
Fecal Incontinence Quality of life Score | 24 months
  Change in quality of life score measured on a scale between 1 and 4, where 1 is very affected and 4 is not affected
Resting pressure (mm hg) | 3 months
  Pressure during relaxation of the anal sphincter
Squeeze pressure (mm hg) | 3 months
  Pressure during contraction of the anal sphincter
First sensation (volume of the balloon by cm water) | 3 months
  First sensation of the stool in the rectum
First Urge (volume of the balloon by cm water) | 3 months
  The patient is trying to hold defecation and he can

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Kharoub, MD, Study Director — faculty of medicine, Benha university
Locations (1):
- Benha University, Banhā, Al Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After Publication, investigators would like to share the data with other researchers who interested in this topic
Supporting Information: Study Protocol
Time Frame: After Publication
Access Criteria: Not available now